CLINICAL TRIAL: NCT04886973
Title: Effect of Insulin Resistance on Branched Chain Amino Acid Metabolism.
Acronym: BCAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Maria Viridiana Olin Sandoval, Medical Sciences Investigator C, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FNU-3549-20-23-1
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with a Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) ≥ 2.5 (Experimental): Administration of an 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids. The dose will be calculated considering the 25% of the estimated protein per day (1 g/kg/day). This dose will be placed in a short peripheral intravenous catheter and administered at a rate of 1.5ml per minute, using an infusion pump. The patient will be monitored all the time by a physician.
  Interventions: Other: Administration of an 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids.
- Subjects with a Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) < 2.5 (Experimental): Administration of an 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids. The dose will be calculated considering the 25% of the estimated protein per day (1 g/kg/day). This dose will be placed in a short peripheral intravenous catheter and administered at a rate of 1.5ml per minute, using an infusion pump. The patient will be monitored all the time by a physician.
  Interventions: Other: Administration of an 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids.

INTERVENTIONS:
Other: Administration of an 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids. — Intravenous administration of 8% crystalline L-amino acids with high concentrations of branched chain amino acids.

SUMMARY:
It has been observed that subjects with obesity and insulin resistance have higher concentrations of branched chain amino acids in plasma or serum. However, this association has been established under fasting conditions, so they only give information about a metabolic state and do not reflect the dynamics and flexibility of the metabolism of these amino acids in the absence or presence of insulin resistance. The main aim of this study is to compare the catabolism of branched chain amino acids and their keto acids in subjects with and without insulin resistance, after the infusion of an amino acid solution with high concentration of the branched chain amino acids, leucine, valine, and isoleucine. The results of this project will allow the investigators to understand the dynamics of the branched chain amino acids and their derivatives, and its relationship with insulin resistance, which could eventually be used to design nutritional strategies to treat insulin resistance and thus, delay the development of type 2 diabetes.

DETAILED DESCRIPTION:
An 8% crystalline L-amino acid solution with high concentrations of branched chain amino acids, leucine, isoleucine, and valine, will be administered intravenously. The dose will be calculated considering the 25% of the estimated protein per day. For example, if the patient is 70 kg and the investigators consider 1g/kg/day, the amount of protein to be administered will be 17.5 grams (70 x 0.25 = 17.5 grams). This dose will be placed in a short peripheral intravenous catheter and administered at a rate of 1.5ml per minute, using an infusion pump. The patient will be monitored all the time by a physician. After the administration of the L- amino acid solution, the investigators will take blood samples at 0, 15, 30, 45, 60, 90 and 120 minutes to determine the area under the curve for glucose, insulin, amino acids and branched chain keto acids.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for cases (subjects with insulin resistance).

* Male and female.
* Adults between 18 and 50 years of age.
* Body Mass Index (BMI) ≥ 18.5 and ≤ 40 kg/m2.
* HOMA index ≥ 2.5
* In the case of women, being in the follicular phase of the menstrual cycle.

Inclusion criteria for controls (subjects without insulin resistance).

* Male and female
* Adults between 18 and 50 years of age.
* Body Mass Index (BMI) ≥ 18.5 and ≤ 40 kg/m2.
* HOMA index < 2.5
* Blood glucose < 100 mg/dL
* In the case of women, being in the follicular phase of the menstrual cycle.

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with kidney disease diagnosed by any physician.
* Patients with creatinine > 1.3 mg/dL for men and > 1.1 mg/dL for women and/or Blood Urea Nitrogen (BUN) > 20 mg/dL.
* Patients with acquired diseases secondarily producing obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Weight loss > 3 kg in the last 3 months.
* Patients with any catabolic diseases.
* Pregnancy status.
* Positive smoking.
* Treatment with any medication (except contraceptives and proton pump inhibitors)
* Having suffered any infection in the last 20 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Area under the curve of branched-chain amino acids. | 2 hours
  Time Frame: Measured for 0,15,30,45,60,90,120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The branched chain amino acids concentration will be determined by liquid chromatography coupled to mass spectrometry (LC-MS/MS), and the area under the curve will be calculated using the trapezoidal rule.

SECONDARY OUTCOMES:
Area under the curve of branched-chain keto acids. | 2 hours
  Time Frame: Measured for 0,15,30,45,60,90,120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The branched chain keto acids concentration will be determined by liquid chromatography coupled to mass spectrometry (LC-MS/MS), and the area under the curve will be calculated using the trapezoidal rule.
Area under the curve of insulin. | 2 hours
  Time Frame: Measured for 0,15,30,45,60,90,120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The insulin concentration will be determined using an ELISA assay and the area under the curve will be calculated using the trapezoidal rule.
Area under the curve of glucose. | 2 hours
  Time Frame: Measured for 0,15,30,45,60,90,120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The glucose concentration will be determined using an enzymatic assay (Hexokinase) and the area under the curve will be calculated using the trapezoidal rule.
Respiratory quotient. | 2 hours
  Time Frame: Measured for 0,15,30,45,60,90,120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids The respiratory quotient will be determined by indirect calorimetry and the area under the curve will be calculated using the trapezoidal rule.
Expression of the enzyme branched-chain aminotransferase 2 (BCAT2) | 2 hours
  Time Frame: Measured for 0, 60 and 120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The expression of enzyme branched chain aminotransferase 2 (BCAT2) will be determined in mononuclear cells isolated from blood by Western Blot and quantitative PCR.
Expression of the enzyme branched-chain keto acid dehydrogenase (BCKDH) | 2 hours
  Time Frame: Measured for 0, 60 and 120 minutes following the intravenous administration of the amino acid solution rich in branched chain amino acids.
  The expression of enzyme branched chain ketoacid dehydrogenase (BCKDH) will be determined in mononuclear cells isolated from blood by Western Blot and quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA VIRIDIANA OLIN SANDOVAL, Dr, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas Y Nutricion Salvador Zubiran, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shimomura Y, Yamamoto Y, Bajotto G, Sato J, Murakami T, Shimomura N, Kobayashi H, Mawatari K. Nutraceutical effects of branched-chain amino acids on skeletal muscle. J Nutr. 2006 Feb;136(2):529S-532S. doi: 10.1093/jn/136.2.529S. PMID 16424141
- [Background] Zhang S, Zeng X, Ren M, Mao X, Qiao S. Novel metabolic and physiological functions of branched chain amino acids: a review. J Anim Sci Biotechnol. 2017 Jan 23;8:10. doi: 10.1186/s40104-016-0139-z. eCollection 2017. PMID 28127425
- [Background] Brosnan JT, Brosnan ME. Branched-chain amino acids: enzyme and substrate regulation. J Nutr. 2006 Jan;136(1 Suppl):207S-11S. doi: 10.1093/jn/136.1.207S. PMID 16365084
- [Background] Newgard CB, An J, Bain JR, Muehlbauer MJ, Stevens RD, Lien LF, Haqq AM, Shah SH, Arlotto M, Slentz CA, Rochon J, Gallup D, Ilkayeva O, Wenner BR, Yancy WS Jr, Eisenson H, Musante G, Surwit RS, Millington DS, Butler MD, Svetkey LP. A branched-chain amino acid-related metabolic signature that differentiates obese and lean humans and contributes to insulin resistance. Cell Metab. 2009 Apr;9(4):311-26. doi: 10.1016/j.cmet.2009.02.002. PMID 19356713
- [Background] Floegel A, Stefan N, Yu Z, Muhlenbruch K, Drogan D, Joost HG, Fritsche A, Haring HU, Hrabe de Angelis M, Peters A, Roden M, Prehn C, Wang-Sattler R, Illig T, Schulze MB, Adamski J, Boeing H, Pischon T. Identification of serum metabolites associated with risk of type 2 diabetes using a targeted metabolomic approach. Diabetes. 2013 Feb;62(2):639-48. doi: 10.2337/db12-0495. Epub 2012 Oct 4. PMID 23043162
- [Background] Zhao X, Han Q, Liu Y, Sun C, Gang X, Wang G. The Relationship between Branched-Chain Amino Acid Related Metabolomic Signature and Insulin Resistance: A Systematic Review. J Diabetes Res. 2016;2016:2794591. doi: 10.1155/2016/2794591. Epub 2016 Aug 25. PMID 27642608
- [Background] Wang TJ, Larson MG, Vasan RS, Cheng S, Rhee EP, McCabe E, Lewis GD, Fox CS, Jacques PF, Fernandez C, O'Donnell CJ, Carr SA, Mootha VK, Florez JC, Souza A, Melander O, Clish CB, Gerszten RE. Metabolite profiles and the risk of developing diabetes. Nat Med. 2011 Apr;17(4):448-53. doi: 10.1038/nm.2307. Epub 2011 Mar 20. PMID 21423183
- [Background] Lynch CJ, Adams SH. Branched-chain amino acids in metabolic signalling and insulin resistance. Nat Rev Endocrinol. 2014 Dec;10(12):723-36. doi: 10.1038/nrendo.2014.171. Epub 2014 Oct 7. PMID 25287287
- [Background] Serralde-Zuniga AE, Guevara-Cruz M, Tovar AR, Herrera-Hernandez MF, Noriega LG, Granados O, Torres N. Omental adipose tissue gene expression, gene variants, branched-chain amino acids, and their relationship with metabolic syndrome and insulin resistance in humans. Genes Nutr. 2014 Nov;9(6):431. doi: 10.1007/s12263-014-0431-5. Epub 2014 Sep 27. PMID 25260659
- [Background] Gunnerud U, Holst JJ, Ostman E, Bjorck I. The glycemic, insulinemic and plasma amino acid responses to equi-carbohydrate milk meals, a pilot- study of bovine and human milk. Nutr J. 2012 Oct 12;11:83. doi: 10.1186/1475-2891-11-83. PMID 23057765